CLINICAL TRIAL: NCT06740019
Title: A Phase Ib, Open Label, Multicenter Clinical Study to Evaluate the Safety, Tolerance, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of JMKX000197 Injection in the Treatment of Malignant Pleural Effusion
Brief Title: A Phase Ib Study of JMKX000197 Injection in the Treatment of Malignant Pleural Effusion
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JY-JM-0197-102
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-12

CONDITIONS: Malignant Pleural Effusions (Mpe)
MeSH Terms: conditions — Pleural Effusion, Malignant; Myeloproliferative Disorder, Chronic, with Eosinophilia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (Experimental): JMKX000197 Dose 1
  Interventions: Drug: JMKX000197
- Arm B (Experimental): JMKX000197 Dose 2
  Interventions: Drug: JMKX000197
- Arm C (Other): Tube thoracostomy drainage
  Interventions: Procedure: Tube thoracostomy drainage

INTERVENTIONS:
Drug: JMKX000197 — for pleural perfusion
  Arms: Arm A; Arm B
Procedure: Tube thoracostomy drainage — Tube thoracostomy drainage
  Arms: Arm C

SUMMARY:
A Phase Ib Study to Evaluate the Safety, Tolerance, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of JMKX000197 Injection in the Treatment of Malignant Pleural Effusion

ELIGIBILITY:
Inclusion Criteria:

1. The participant voluntarily joined the study, signed an informed consent form, and had good compliance.
2. Age ≥ 18 years and ≤ 75 years old, regardless of gender.
3. Participants with advanced solid tumors diagnosed by histopathology or cytopathology.
4. Malignant pleural effusion confirmed by histopathology or cytopathology or clinically diagnosed as moderate or above and requiring drainage.
5. Eastern Cooperative Oncology Group (ECOG) performance status: 0 to 2.
6. Life expectancy of at least 3 months.
7. Adequate organ function.
8. Female participants of childbearing potential should agree to use contraception to prevent pregnancy until 6 months after discontinuation of JMKX000197. The serum pregnancy test result should be negative 7 days before enrollment and must be a non-lactating participant. Male participants must agree to use effective contraception during the study and for 6 months after discontinuation of JMKX000197.

Exclusion Criteria:

1. Bilateral pleural effusion or concurrent peritoneal effusion, or concurrent pericardial effusion.
2. Pleural effusion is either encapsulated or severely separated; Or merge with chylothorax; Or combined with infectious pleural effusion.
3. Have used interferon gene stimulating factor (STING) agonists for pleural perfusion。
4. Known allergies to the study drug or its excipient components.
5. Have participated in other clinical trials within 28 days prior to randomization.
6. Major surgery within 28 days prior to randomization.
7. Central nervous system metastatic disease, leptomeningeal disease, or cord compression.
8. Clinical unstable or uncontrolled concomitant cardiovascular, pulmonary, hepatic, renal or seizures diseases.
9. Uncontrollable systemic infections (viruses, bacteria, fungi), including but not limited to positive HBsAg and HBV DNA, positive HCV RNA, positive HIV antibody test or combined infections within the first 28 days of randomization and require systemic anti-infective treatment.
10. Have a history of organ transplantation.
11. Any further condition which, in the opinion of the Investigator, the participant is not suitable in the present study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
AEs or SAEs | Up to approximately 36 days
Recommended Phase II dose (RP2D) | Up to approximately 24 months

SECONDARY OUTCOMES:
Puncture /drainage-Free Survival (PuFS) | Up to approximately 24 months
Pleural effusion overall response (ORR) | Up to approximately 24 months
Overall survival (OS) | Up to approximately 24 months
Pharmacokinetics (Cmax) | Up to approximately 7 days
Pharmacokinetics(Tmax) | Up to approximately 7 days
Pharmacokinetics (t1/2) | Up to approximately 7 days
Pharmacokinetics (AUC0-inf) | Up to approximately 7 days
Pharmacokinetics (AUC0-t) | Up to approximately 7 days
Amount of Drug Excreted Via Urine and Excrement | Up to approximately 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No